CLINICAL TRIAL: NCT03590171
Title: International Study for Treatment of High Risk Childhood Relapsed ALL 2010 A Randomized Phase II Study Conducted by the Resistant Disease Committee of the International Berlin, Frankfurt, Münster (BFM) Study Group
Brief Title: International Study for Treatment of High Risk Childhood Relapsed ALL 2010
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Australian & New Zealand Children's Haematology/Oncology Group (Other); St. Anna Kinderkrebsforschung, CCRI (co-sponsor, Austria) (Unknown); European Organisation for Research and Treatment of Cancer - EORTC (Network); University Hospital, Motol (Other); Rigshospitalet, Denmark (Other); Turku University Central Hospital (co-sponsor, Finland) (Unknown); Centre Hospitalier Universitaire de Nice (Other); Our Lady's Chilrden's Hospital (Co-Sponsor Ireland) (Unknown); Tel Aviv Sourasky Medical Centre (Co-Sponsor Israel) (Unknown); Ospedale Pediatrico Bambino (co-sponsor, Italy) (Unknown); Prinses Máxima Centrum (Co-Sponsor Netherlands) (Unknown); Oslo University Hospital (co-sponsor, Norway) (Unknown); Medical University of Wroclaw (Co-Sponsor Poland) (Unknown); Instituto Português de Oncologia de Lisboa (co-sponsor, Portugal) (Unknown); Karolinska University Hospital Stockholm (co-sponsor, Sweden) (Unknown); Spanish Society of Pediatric Hematology and Oncology (SEHOP) (Co-Sponsor Spain) (Unknown); University Children's Hospital, Zurich (Other); Central Manchester University Hospitals NHS Foundation Trust (co-sponsor, UK) (Unknown)
Responsible Party: Principal Investigator, PD Dr. Arend von Stackelberg, Prinicipal Investigator, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IntReALL HR 2010
Record Dates: First submitted 2018-05-23; First posted 2018-07-18 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Acute Lymphoblastic Leukemia (ALL)
Keywords: ALL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm HR-A (No Intervention): Induction: Backbone ALL R3
- Arm HR-B (Experimental): Induction: Backbone ALL R3 + Bortezomib
  Interventions: Drug: Bortezomib

INTERVENTIONS:
Drug: Bortezomib — Patients randomised to the HR-B arm receive induction, consolidation with the modified ALL R3 protocol. In this arm, patients are randomized to receive Bortezomib together with the ALL R3 protocol during induction. Administration of Bortezomib: 1.3 mg/m2 as intravenous bolus or subcutaneously (SC, at the discretion of the treating physician) on days 1 and 4 of weeks 1 and 3.
  Arms: Arm HR-B

SUMMARY:
The main goal of this study is to improve the outcome of children and adolescents with acute lymphoblastic leukemia with high risk first relapse by optimization of treatment strategies within a large international trial and the integration of new agents.

DETAILED DESCRIPTION:
Though survival of children with acute lymphoblastic leukemia (ALL) has considerably improved over the past few decades, relapsed ALL remains a leading cause of mortality in children with cancer. Risk has been defined by the International (I) Berlin, Frankfurt, Münster (BFM) Study Group (SG) based on duration of first remission, immunophenotype of malignant clone, and site of relapse. Patients classified as high risk (HR) by these criteria have poor response rates to standard induction therapy, high rates of subsequent relapse and require an allogeneic hematopoetic stem cell transplantation (allo-HSCT) for consolidation of 2nd remission. Over the last decade members of the I-BFM-SG have investigated the use of different combinations of conventional cytotoxic agents. Even with allo-HSCT, none of these approaches have improved outcome above 40%. Therefore, for HR patients there is a need to investigate the curative potential of new agents combined with systemic therapy. The proteasome inhibitor bortezomib has shown synergistic activity with acceptable toxicity when combined with corticosteroids, anthracyclines and alkylating agents in adult patients with cancer as well as with dexamethasone, doxorubicin, vincristine and polyethylene glycol (PEG) asparaginase in children with refractory or relapsed ALL. In the I-BFM-SG International Study for Treatment of High Risk Childhood Relapsed ALL (IntReALL) HR 2010 study, the potential of Bortezomib combined with a modified ALL relapse protocol 3 (R3) backbone as induction regimen for HR patients to improve complete 2nd remission (CR2) rates will be investigated in a randomized phase II design. Induction is followed by conventional intensive consolidation. After termination of the trial patients may be subjected to an investigational window, before all of them receive allo-HSCT.

ELIGIBILITY:
Inclusion Criteria:

* Morphologically confirmed diagnosis of 1st relapsed precursor B-cell or T-cell ALL
* Children less than 18 years of age at date of inclusion into the study
* Meeting HR criteria any BM relapse, early/very early isolated BM relapse, very early isolated/combined extramedullary relapse)
* Patient enrolled in a participating centre
* Written informed consent
* Start of treatment falling into the study period
* No participation in other clinical trials 30 day prior to study enrolment that interfere with this protocol, except trials for primary ALL

Exclusion Criteria:

* Breakpoint cluster region-Abelson (BCR-ABL)/ t(9;22) positive ALL
* Pregnancy or positive pregnancy test (urine sample positive for β-humane choriongonadotropin (HCG) > 10 U/l)
* Sexually active adolescents not willing to use highly effective contraceptive method (pearl index <1) until 12 months after end of anti-leukemic therapy
* Breast feeding
* Relapse post allogeneic stem-cell transplantation
* Neuropathy > II°
* The whole protocol or essential parts are declined either by patient himself/herself or the respective legal guardian
* Objection to the study participation by a minor patient, able to object
* Any patient being dependent on the investigator
* No consent is given for saving and propagation of pseudonymized medical data for study reasons
* Severe concomitant disease that does not allow treatment according to the protocol at the investigator's discretion (e.g. malformation syndromes, cardiac malformations, metabolic disorders)
* Subjects unwilling or unable to comply with the study procedures
* Subjects who are legally detained in an official institute

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 250 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of Complete Remission | Week 4
  Rate of complete second remission (CR2) quantified by cytology after induction with standard chemotherapy + bortezomib (arm B) compared with standard chemotherapy (arm A).

SECONDARY OUTCOMES:
Event-free Survival | Year 3
  Improvement of three years event-free survival (EFS)
Overall Survival | Year 3
  Improvement of three years overall survival (OS)
Minimal Residual Disease Reduction (MRD) | Week 4
  Improvement of Minimal Residual Disease (MRD) reduction after induction with versus without bortezomib
Minimal Residual Disease Load | Week 15
  Improvement of MRD load prior to stem cell transplantation (SCT).
Minimal Residual Disease (MRD) | Week 15
  Prognostic relevance of MRD pre stem cell transplantation (SCT). MRD will be quantified before stem cell transplantation with polymerase chain reaction (PCR) and will be related to EFS after SCT. Multicolour flow cytometry will be used in parallel with PCR. Flow cytometry is used instead of PCR if PCR based MRD-quantification cannot be performed, because criteria for a reliable and reproducible sensitive quantification are not fulfilled.
Complete Remission/Minimal Residual Disease Rates During Consolidation | Week 5, 8, 11, 15
  Improvement of CR2 and/or MRD rates during consolidation
Toxicity of induction classified with the COMMON TOXICITY CRITERIA (CTC) | At induction up to week 5
  Toxicity of induction with versus without bortezomib. Toxicity of the central nervous system and peripheral neuropathy will be classified with the COMMON TOXICITY CRITERIA (CTC).

OTHER OUTCOMES:
Minimal Residual Disease in Isolated Extramedullary Relapse | Day 0; Week 5, 8, 11, 15
  The rate and extent of sub-microscopic bone marrow (BM) involvement in extramedullary leukemia will be investigated prospectively.
Extended Genetic Characterization | Day 0
  Extension of genetic characterization and correlation with clinical data
In-vitro drug response profile | Day 0
  Generation of primografts from patient samples for bio-banking and drug testing by using immunodeficient mice. The outcome measure is the in-vitro drug response profile using the primograft of primary patient sample. The in-vitro drug response profile will be compared to the in-vivo drug response of a patient. In order to get an "in-vitro drug response profile" apoptosis/viability of the primary patient sample or patient-derived xenograft sample is measured using different concentrations of novel drugs normally after 48 hours of treatment. These drugs could be potentially given to a patient, when there will be no response to conventional protocol treatment. Apoptosis/viability is measured by live cell imaging microscopy or/and by flow cytometry. The report will include half maximal inhibitory concentration (IC50), the concentration of a drug which kills half of the cell after a defined time (normally 48h) for a variety of potential drugs.

CONTACTS AND LOCATIONS:
Overall Officials: Arend von Stackelberg, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (15):
- Australian & New Zealand Childhood Hematology & Oncology Group, Clayton, Victoria, Australia
- St. Anna Kinderkrebsforschung, CCRI, Vienna, Austria
- Hòpital Universitaire des Enfants Reine Fabiola, Brussels, Belgium
- University Hospital Motol, Prague, Czechia
- Copenhagen University Hospital (Rigshospitalet), Copenhagen, Denmark
- Turku University Central Hospital, Turku, Finland
- CHU Nice, Nice, France
- Tel Aviv Sourasky Medical Centre, Tel Aviv, Israel
- Ospedale Pediatrico Bambino Gesù, Roma, Italy
- Prinses Máxima Centrum, Lundlaan, Utrecht, Netherlands
- Oslo University Hospital, Oslo, Norway
- Dpt. SCT and Hematology/Oncology University Wroclaw, Wroclaw, Poland
- Instituto Português de Oncologia de Lisboa, Lisbon, Portugal
- University Hospital Stockholm, Stockholm, Sweden
- Royal Manchester Children's Hospital, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided